CLINICAL TRIAL: NCT04542512
Title: Risk Factors for Necrotic Cholecystitis During COVID-19 Pandemic: the ChoCO-WSES Prospective Observational Multicenter International Study.
Brief Title: Risk Factors for Necrotic Cholecystitis During COVID-19 Pandemic.
Acronym: ChoCO-W
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poissy-Saint Germain Hospital (Other)
Collaborators: World Society of Emergency Surgery (Other); Intercontinental society of Natural Orifice, Endoscopic, and Laparoscopic Surgery (Unknown)
Responsible Party: Principal Investigator, Belinda De Simone, General Surgeon, Poissy-Saint Germain Hospital
Other Study IDs: 06012020
Record Dates: First submitted 2020-09-06; First posted 2020-09-09 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Cholecystitis, Acute; Cholecystitis; Gangrenous; Cholecystitis Suppurative; Covid19
Keywords: COVID-19; emergency surgery; acute abdomen; peritonitis; cholecystitis; necrotic cholecystitis; percutaneous drainage of gallbladder; laparoscopic cholecystectomy; operative management; timing of cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis; Gangrene; COVID-19; Abdomen, Acute; Peritonitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gangrenous cholecystitis is the most common complication of acute cholecystitis.

Preliminary data showed that COVID-19 patients have a high risk to present necrotic cholecystitis.

The Cholecystitis under COVID-19 pandemic WSES (ChoCO-W) study aims to investigate risk factors and high-risk patients to develop necrotic cholecystitis during this pandemic and their management.

DETAILED DESCRIPTION:
Background:

Gangrenous cholecystitis is the most common complication of acute cholecystitis affecting around 15% (range 2-30%) of patients and it occurs as a result of ischemia with necrosis of the gallbladder wall [1].

It is related to an increased mortality rate (mortality rate ranging between 15 and 50%) compared with non-necrotic acute cholecystitis[2].

Retrospective studies that investigated risk and predictive factors related to gangrenous cholecystitis showed that males, older patients with diabetes, coronary artery disease, and other comorbidities are at risk to present with gangrenous cholecystitis. [1-3] Another study identified longer delay time prior to hospital admission and low white blood cell count as independent risk factors affecting mortality and indicated the presence of diabetes mellitus, higher blood levels of aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase and total bilirubin, pericholecystic fluid in abdominal ultrasonography, and conversion from laparoscopic surgery to open surgery as risk factors increasing mortality [2] In any case, the treatment of GC is similar to that of patients with AC but in the presence of GC, cholecystectomy can be difficult because of adhesions, insufficient anatomic control, complications like bleeding, and injury to bile ducts.

There is high variability in the reported conversion rate to be 30% to 50% [4], down to 8.7% [5]. These results are probably due to a careful preoperative selection of patients for laparoscopic cholecystectomy and early surgery [6].

Hunt et al [7] reported decreased morbidity and mortality rates with the implementation of laparoscopic cholecystectomy for GC.

Onder et al [2] showed that mortality was higher in cases in which conversion to open surgery occurred.

Recently, many authors reported necrotic and perforated cholecystitis as the most common complication of COVID-19 pneumonia [8-9-10].

A recent multi-society position paper suggested to consider percutaneous drainage of the gallbladder after the failure of conservative therapy with antibiotics but highlighted that advanced age, or other factors of higher COVID-19 risk, cannot be regarded as sufficient to indicate this alternative treatment except in real conditions of the impracticability of cholecystectomy [11].

In the lack of evidence and guidelines about the management of a patient with acute cholecystitis during COVID-19 pandemic, laparoscopic cholecystectomy, at most preceded by percutaneous trans-gallbladder drainage (PTGBD) in high surgical risk patients, remains the gold standard for the treatment of acute cholecystitis on COVID-19 patients, with high morbidity rate and length of hospital stay that increases the risk of spreading the virus among health care staff and negative COVID-19 patients.

The study aims to evaluate the incidence and mortality of necrotic cholecystitis among Covid (+) patients under the COVID-19 pandemic, to improve their management and to confirm that COVID-19 infection is a risk factor for necrotic cholecystitis; to assess the management of acute cholecystitis during COVID-19 pandemic.

The rationale for the trial:

* Investigate the risk factors to develop necrotic cholecystitis under the COVID-19 pandemic;
* Evaluate the management of acute cholecystitis focusing on treatments and outcomes of the operative or non-operative management in COVID (+) and COVID (-) patients to improve outcomes, decreasing morbidity and mortality rates related to emergency setting and high-risk patients;
* Confirm that COVID-19 disease is a risk factor for necrotic cholecystitis.

Objectives:

Evaluate the incidence of necrotic cholecystitis during the COVID-19 pandemic among Covid patients; Evaluate the prevalence of necrotic cholecystitis in patients presenting with acute cholecystitis during the COVID-19 pandemic; Evaluate the risk factors for necrotic cholecystitis in COVID-19 patients and negative ones.

Confirm the hypothesis that COVID-19 infection is a risk factor for necrotic cholecystitis; Evaluate the clinical outcomes of early (<72h from the onset of symptoms) versus delayed (>72h from the onset of symptoms) cholecystectomy, and of a non operative management according to the WSES international guidelines (2020) for the management of calculus cholecystitis and Tokyo severity classification for cholecystitis, in terms of mortality and morbidity.

Primary endpoints To evaluate the prevalence of necrotic cholecystitis among patients admitted for acute cholecystitis during the Covid-19 pandemic; The incidence of necrotizing cholecystitis in the cohort of COVID-19 positive patients; To assess mortality due to necrotic cholecystitis during the Covid-19 pandemic among Covid-19 infected patients

Secondary endpoints To investigate the risk factors for necrotic cholecystitis in patients admitted with diagnosis of acute cholecystitis and in the cohort of Covid-19 patients; to investigate if the COVID-19 infection is a risk factor to present necrotic cholecystitis; to assess the management of acute cholecystitis during Covid-19 pandemic and the role of non operative management strategy and operative management.

Study Design:

International Observational Prospective Cohort Study.

Study population:

All adult patients admitted to the surgical department with a diagnosis of acute cholecystitis (with and without necrotising cholecystitis).

Inclusion criteria Patients of all age and sex admitted in the emergency department for acute cholecystitis, aged >=18 years old.

Exclusion criteria Patients aged< 18 years old.

Period April 2021-September 2021

Data collection All epidemiological, clinical, surgical and follow up data will be collected on an online case report form.

Sample size calculation This is an explorative study and data will be used to investigate risk factors, prevalence of necrotic cholecystitis among patients admitted with diagnosis of acute cholecystitis during COVID-19 pandemic, and the specific characteristics behind the choice between early cholecystectomy, delayed cholecystectomy, radiological drainage of the gallbladder and medical treatment (antibiotics) in an emergency setting.

We calculated the sample size by considering the incidence of necrotic cholecystitis reported in literature which corresponds to a range of 2-30%. Taking into account the mean between the 2 values, and in the lack of data on the incidence of necrotic cholecystitis in Covid patients, that we assumed to be double the incidence of necrotic cholecystitis in non-Covid population, with an alfa risk estimated error equal to 0.05, the study population will be composed of 2 cohorts of 111 patients

Statistical analysis This is a study evaluating the prevalence of necrotic cholecystitis among patients admitted for acute cholecystitis during COVID-19 pandemic and the incidence of necrotic cholecystitis in Covid (+) patients. An univariate and multivariate analysis of each scheduled parameter will be carried out. In the statistical analysis, the investigator will differentiate data by cohorts (Covid (-) and Covid (+) patients) and gender. The main aim of this study is to assess the management of all patients having acute cholecystitis during COVID-19.

Primary endpoints:

In hospital mortality among patients with acute necrotic cholecystitis In hospital mortality among Covid-19 patients presenting with acute necrotic cholecystitis

Secondary endpoints To assess the risk factors for necrotic cholecystitis in Covid+ patients; To evaluate the management of acute cholecystitis during the Covid-19 pandemic (medical treatment, surgical treatment, medical treatment and radiological drainage of the gallbladder); To confirm that COVID-19 infection is a risk factor for developing necrotic cholecystitis.

Ethical Aspects This is an observational study. It will not attempt to change or modify the clinical practice of the participating physicians. All surgeons involved in the patient's recruitment will be included in the research authorship. This is an observational study, it will not attempt to change or modify the clinical practice of the participating physicians. The study will meet and conform to the standards outlined in the Declaration of Helsinki and Good Epidemiological Practices.

Every clinical centre attending the study is responsible for Ethics Committee approval.

All surgeons involved in the patients' recruitment will be included in the research authorship.

Methods and assessments:

Every clinical centre will be identified by a number assigned by the principal investigator before starting data entry. An online case report form will be available to collect data: the link for the access will be sent to the local investigator, to share with local collaborators.

Safety Considerations There are no safety issues

Informed consent This observational study will not attempt to change or modify the laboratory or clinical practices of the participating physicians, consequently informed consent will not be required. Each eligible patient for this study will be asked to sign a written consent to authorize the anonymous treatment of personal data, according to standard clinical practice.

Data Management and Statistical Analysis Every local investigator is responsible for data entry. Prof. Fikri Abu-Zidan is the coordinator of statistical analysis.

Expected Outcomes of the Study The aim of this study is to demonstrate the the correlation between necrotic cholecystitis and predisposition to thrombo-embolism in COVID-19 patients and that the patients presenting one or more risk factors for necrotic cholecystitis have to be managed operatively without long delay if fit for surgery.

Dissemination of Results and Publication Policy The primary outcomes of the study will be presented at the World Congress of the World Society of Emergency Surgery in September 2021. The ChoCO-W study embraces corporate authorship and all collaborators that contribute to this study will form the ChoCO-W collaborative group. This group will co-author all publications in which ChoCO-W study data is used.

Duration of the Project 2 years

Ethics This is an observational study.

Budget No budget study

Financing and Insurance Not applicable

ELIGIBILITY:
Inclusion Criteria:

All patients presenting acute cholecystitis during COVID 19 pandemic, aged >=18 yo

Exclusion Criteria:

Patients presenting with acute cholecystitis aged <18 yo

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the surgical department with clinical and histologic diagnosis of acute cholecystitis (with and without gangrenous cholecystitis).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between COVID-19 pneumonia and necrotic cholecystitis | through study completion, an average of 1 year
  Incidence of necrotic cholecystitis in COVID-19 patients
Correlation between coagulopathy and necrotic cholecystitis | through study completion, an average of 1 year
  mortality related to necrotising cholecystitis in COVID-19 patients
Outcome necrotic cholecystitis during COVID-19 pandemic | through study completion, an average of 1 year
  overall mortality

SECONDARY OUTCOMES:
Correlation between coagulopathy and necrotic cholecystitis | through study completion, an average of 1 year
  D-Dimer value
Risk factors for necrotic cholecystitis | through study completion, an average of 1 year
  COVID-19 infection
Correlation between coagulopathy and necrotic cholecystitis | through study completion, an average of 1 year
  Mean INR value
Correlation between coagulopathy and necrotic cholecystitis | through study completion, an average of 1 year
  Mean Prothrombin time (PT; sec); mean activated partial thromboplastin (aPT; sec)
Correlation between coagulopathy and necrotic cholecystitis | through study completion, an average of 1 year
  Mean Fibrinogen value (g/L)
Correlation between coagulopathy and necrotic cholecystitis | through study completion, an average of 1 year
  most common alterations of thromboelastography

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal Poissy-Saint Germain en Laye, Poissy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eldar S, Eitan A, Bickel A, Sabo E, Cohen A, Abrahamson J, Matter I. The impact of patient delay and physician delay on the outcome of laparoscopic cholecystectomy for acute cholecystitis. Am J Surg. 1999 Oct;178(4):303-7. doi: 10.1016/s0002-9610(99)00172-5. PMID 10587188
- [Background] Ying M, Lu B, Pan J, Lu G, Zhou S, Wang D, Li L, Shen J, Shu J; From the COVID-19 Investigating and Research Team. COVID-19 with acute cholecystitis: a case report. BMC Infect Dis. 2020 Jun 22;20(1):437. doi: 10.1186/s12879-020-05164-7. PMID 32571224
- [Background] Bruni A, Garofalo E, Zuccala V, Curro G, Torti C, Navarra G, De Sarro G, Navalesi P, Longhini F, Ammendola M. Histopathological findings in a COVID-19 patient affected by ischemic gangrenous cholecystitis. World J Emerg Surg. 2020 Jul 2;15(1):43. doi: 10.1186/s13017-020-00320-5. PMID 32615987
- [Background] Campanile FC, Podda M, Arezzo A, Botteri E, Sartori A, Guerrieri M, Cassinotti E, Muttillo I, Pisano M, Brachet Contul R, D'Ambrosio G, Cuccurullo D, Bergamini C, Allaix ME, Caracino V, Petz WL, Milone M, Silecchia G, Anania G, Agrusa A, Di Saverio S, Casarano S, Cicala C, Narilli P, Federici S, Carlini M, Paganini A, Bianchi PP, Salaj A, Mazzari A, Meniconi RL, Puzziello A, Terrosu G, De Simone B, Coccolini F, Catena F, Agresta F. Acute cholecystitis during COVID-19 pandemic: a multisocietary position statement. World J Emerg Surg. 2020 Jun 8;15(1):38. doi: 10.1186/s13017-020-00317-0. PMID 32513287
- [Result] Bourikian S, Anand RJ, Aboutanos M, Wolfe LG, Ferrada P. Risk factors for acute gangrenous cholecystitis in emergency general surgery patients. Am J Surg. 2015 Oct;210(4):730-3. doi: 10.1016/j.amjsurg.2015.05.003. Epub 2015 Jun 27. PMID 26186803
- [Result] Onder A, Kapan M, Ulger BV, Oguz A, Turkoglu A, Uslukaya O. Gangrenous cholecystitis: mortality and risk factors. Int Surg. 2015 Feb;100(2):254-60. doi: 10.9738/INTSURG-D-13-00222.1. PMID 25692427
- [Result] Gomes CA, Soares C, Di Saverio S, Sartelli M, de Souza Silva PG, Orlandi AS, Heringer TL, Gomes FC, Catena F. Gangrenous cholecystitis in male patients: A study of prevalence and predictive risk factors. Ann Hepatobiliary Pancreat Surg. 2019 Feb;23(1):34-40. doi: 10.14701/ahbps.2019.23.1.34. Epub 2019 Feb 28. PMID 30863805
- [Result] Contini S, Corradi D, Busi N, Alessandri L, Pezzarossa A, Scarpignato C. Can gangrenous cholecystitis be prevented?: a plea against a "wait and see" attitude. J Clin Gastroenterol. 2004 Sep;38(8):710-6. doi: 10.1097/01.mcg.0000135898.68155.88. PMID 15319657
- [Result] Pisano M, Ceresoli M, Cimbanassi S, Gurusamy K, Coccolini F, Borzellino G, Costa G, Allievi N, Amato B, Boerma D, Calcagno P, Campanati L, Campanile FC, Casati A, Chiara O, Crucitti A, di Saverio S, Filauro M, Gabrielli F, Guttadauro A, Kluger Y, Magnone S, Merli C, Poiasina E, Puzziello A, Sartelli M, Catena F, Ansaloni L. 2017 WSES and SICG guidelines on acute calcolous cholecystitis in elderly population. World J Emerg Surg. 2019 Mar 4;14:10. doi: 10.1186/s13017-019-0224-7. eCollection 2019. PMID 30867674
- [Result] Hunt DR, Chu FC. Gangrenous cholecystitis in the laparoscopic era. Aust N Z J Surg. 2000 Jun;70(6):428-30. doi: 10.1046/j.1440-1622.2000.01851.x. PMID 10843398
- See also: Registration form to collaborate — https://docs.google.com/forms/d/e/1FAIpQLSeu2gIILNlYRHvSa815PSKXWR4Ow2LnXG87vtoujuaP5XwaGg/viewform?usp=sf_link
- See also: Online case report form — https://docs.google.com/forms/d/e/1FAIpQLSfrHWCdiEbo91y1JbHgEtKR9nGR1FWtjiv5RiHJZJe4_ElJ2A/viewform?usp=sf_link